CLINICAL TRIAL: NCT05131269
Title: The Level of Matrix Metalloproteinase-1 (MMP-1), Tissue Inhibitor Matrix Metalloproteinase-1 (TIMP-1) After Prolotherapy Intervention and The Functional Outcome in Patient With Frozen Shoulder
Brief Title: Prolotherapy Intervention in Patient With Frozen Shoulder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bumi Herman (Other)
Responsible Party: Sponsor-Investigator, Bumi Herman, Assistant Lecturer, Hasanuddin University
Organization: Hasanuddin University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0411211741
Record Dates: First submitted 2021-11-04; First posted 2021-11-23 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Frozen Shoulder
Keywords: MMP-1; TIMP-1; Prolotherapy; Functional Outcome; Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Glucose; Water; Prolotherapy; Saline Solution; Injections

STUDY DESIGN:
Intervention Model Description: This study involves two arms assigned randomly for receiving different treatments. One arm for Prolotherapy and Normal Saline in the comparison group.
Masking Description: A sealed envelope of the randomized sequence was given to the investigator and care provider, and participants were recruited consecutively according to the permutation sequence. Participants were masked from the therapy by receiving treatment individually in different rooms and occasions. On the day of the assessment, the physician and laboratory technicians were blinded from group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolotherapy (Experimental): A solution of 7.5 ml of 15% dextrose with 2 ml of 40% lidocaine and 10.5 water is given to these shoulder segments as follows.
  1. Supraspinatus muscle 2-4 ml
  2. Infraspinatus muscle 2-4 ml
  3. Teres minor muscle 2-3 ml,
  4. Subscapularis muscle 2-3 ml.
  5. Intraarticular glenohumeral joint 5 ml
  6. Bursa sub acromial 1-2 ml,
  7. Long head tendon biceps 1-2 ml
  8. Acromioclavicular joint 1 ml
  Interventions: Drug: Dextrose 15 % in Water
- Normal Saline 0.9% (Placebo Comparator): A solution of 20 ml normal saline 0.9% is given to these shoulder segments as follows.
  1. Supraspinatus muscle 2-4 ml
  2. Infraspinatus muscle 2-4 ml
  3. Teres minor muscle 2-3 ml,
  4. Subscapularis muscle 2-3 ml.
  5. Intraarticular glenohumeral joint 5 ml
  6. Bursa sub acromial 1-2 ml,
  7. Long head tendon biceps 1-2 ml
  8. Acromioclavicular joint 1 ml
  Interventions: Drug: Normal Saline 20 mL Injection

INTERVENTIONS:
Drug: Dextrose 15 % in Water — A 15% dextrose solution is given to shoulder segments four times with 2 weeks interval (week 0,2,4, and 6)
  Other Names: Prolotherapy
  Arms: Prolotherapy
Drug: Normal Saline 20 mL Injection — A Normal Saline 0.9% is given to shoulder segments four times with 2 weeks interval (week 0,2,4, and 6)
  Other Names: Comparator
  Arms: Normal Saline 0.9%

SUMMARY:
Introduction :

Prolotherapy is regenerative tissue therapy that is considered to be efficacious in reducing symptoms and morbidity of frozen shoulder, but only a few studies demonstrate the effect of prolotherapy at the biomolecular level, particularly the level of Matrix Metalloproteinase- I (MMP-1), Tissue Inhibitor Matrix Metalloproteinase (TIMP-1), as the biomarkers of cartilage repair.

Objective:

To determine the effect of prolotherapy on MMP-1, TIMP-1, and functional outcomes in frozen shoulder patients

Method:

a double-blind randomized controlled trial study involving participants who had been diagnosed with Frozen Shoulder. History taking, functional outcome assessment, MMP-1, and TIMP-1 were measured. The prolotherapy via intraarticular and extraarticular was performed four times, followed by the evaluation of functional outcome, MMP-1, and TIMP-1 at week 12

Alternative Hypothesis :

Prolotherapy will increase the MMP-1, TIMP-1 levels, and improve functional outcome among Frozen Shoulder patients

DETAILED DESCRIPTION:
Design :

Double-blind randomized trial

Randomization :

Simple Randomization generated by an online randomizer

Sample Size :

Difference between two means of primary outcome where

1. mean difference (μ 1 - μ 2 ) = 0.47
2. pool variance = 0.09
3. Z 1-α/2 = 1.95 with type 1 error 5%
4. 1-β = 1.282 with power 90%. Yielding 16 patients for each arm

Detailed Intervention

1. Intervention group: Prolotherapy is given four times (Week 0, Week 2, Week 4, and Week 6)
2. Comparison group: Normal Saline is given four times with a timeframe similar to the intervention group

Injection location

1. Rotator Cuff muscles
2. Intraarticular glenohumeral joint
3. Subacromial bursa
4. long-heap of the biceps tendon
5. Acromioclavicular joint

Statistical analysis :

1. Descriptive statistic to elaborate baseline characteristic
2. Assuming the baseline characteristic between groups are similar, the independent t-test will be conducted to see the differences between group, whereas Mann Whitney will be performed for nonparametric data
3. Difference within-group (baseline and last day) will be measured by paired-t-test or Wilcoxon for non parametric scenario

ELIGIBILITY:
1. Inclusion Criteria

   1. Age 35-70
   2. Diagnosed with frozen shoulder
   3. At least showing symptoms more than 3 months
2. Exclusion Criteria

   1. Receiving other intraarticular injection
   2. Taking Nonsteroid Antiinflammation drugs 1 week prior to intervention
   3. Skin disorder around the injection site
   4. Septic arthritis

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Matrix Metalloproteinase 1 in Blood | changes of Matrix Metalloproteinase 1 value from baseline to week 6
  Matrix Metalloproteinase 1 from whole blood measured using Enzyme-linked Immunoassay (ELISA). Mean difference between group will be assessed
Tissue Inhibitor Metalloproteinase 1 in Blood | changes of Tissue Inhibitor Metalloproteinase 1 value from baseline to week 6
  Tissue Inhibitor Metalloproteinase 1 from whole blood measured using Enzyme-linked Immunoassay (ELISA). Mean difference between group will be assessed

SECONDARY OUTCOMES:
The Functional Outcome of the Shoulder | changes of Functional Outcome value from baseline to week 6
  The functional outcome is measured using the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire where the patient were asked to do simple task involving the arm, shoulder and hand and also the assessment of additional symptoms and impact to daily life. Higher score indicates disabilities

CONTACTS AND LOCATIONS:
Overall Officials: Nuralam Sarif, MD, Principal Investigator — Hasanuddin University; Irawan Yusuf, PhD, Study Chair — Hasanuddin University; Endy Adnan, PhD, Study Chair — Hasanuddin University; Irfan Idris, PhD, Study Chair — Hasanuddin University
Locations (1):
- Hasanuddin University, Faculty of Medicine, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
De-identified data will be shared accordingly

REFERENCES:
- [Background] Akcay S, Gurel Kandemir N, Kaya T, Dogan N, Eren M. Dextrose Prolotherapy Versus Normal Saline Injection for the Treatment of Lateral Epicondylopathy: A Randomized Controlled Trial. J Altern Complement Med. 2020 Dec;26(12):1159-1168. doi: 10.1089/acm.2020.0286. Epub 2020 Sep 28. PMID 32990454
- [Background] Cho CH, Song KS, Kim BS, Kim DH, Lho YM. Biological Aspect of Pathophysiology for Frozen Shoulder. Biomed Res Int. 2018 May 24;2018:7274517. doi: 10.1155/2018/7274517. eCollection 2018. PMID 29992159
- [Background] Distel LM, Best TM. Prolotherapy: a clinical review of its role in treating chronic musculoskeletal pain. PM R. 2011 Jun;3(6 Suppl 1):S78-81. doi: 10.1016/j.pmrj.2011.04.003. PMID 21703585
- [Background] Lubis AM, Lubis VK. Matrix metalloproteinase, tissue inhibitor of metalloproteinase and transforming growth factor-beta 1 in frozen shoulder, and their changes as response to intensive stretching and supervised neglect exercise. J Orthop Sci. 2013 Jul;18(4):519-27. doi: 10.1007/s00776-013-0387-0. Epub 2013 Apr 19. PMID 23604641
- [Background] Saltzman BM, Leroux T, Meyer MA, Basques BA, Chahal J, Bach BR Jr, Yanke AB, Cole BJ. The Therapeutic Effect of Intra-articular Normal Saline Injections for Knee Osteoarthritis: A Meta-analysis of Evidence Level 1 Studies. Am J Sports Med. 2017 Sep;45(11):2647-2653. doi: 10.1177/0363546516680607. Epub 2016 Dec 27. PMID 28027657